CLINICAL TRIAL: NCT06764446
Title: 6 February 2023 Our Emergency Fasciotomy and Amputation Experiences After Kahramanmaraş Turkey Earthquakes
Brief Title: Our Emergency Fasciotomy and Amputation Experiences
Acronym: Earthquakes
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: Maras Turkey Earthquake
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Amputation; Compartment Syndromes; Earthquake
Keywords: Fasciotomy; Amputation; Earthquakes; 6 February 2023; Kahramanmaraş Turkey Earthquakes; Compartment Syndromes
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Earthquakes are natural disasters that threaten human life and cause loss of life and property in a very short time. In our country, where a large part of the population faces the risk of earthquakes, unfortunately, destructive earthquakes that put the country at a disadvantage in social and economic terms are frequently experienced.

DETAILED DESCRIPTION:
On 6 February 2023, two major earthquakes with a magnitude of 7.7 at 04:17 and 7.6 at 13:24 local time occurred in Kahramanmaraş. In southern Turkey and northern Syria, 11 cities and approximately 14 million people were affected. According to the latest official data, at least 50,783 deaths, more than 122,000 injuries, and major damage occurred. The triage, treatment, and management of the injured was a challenging administrative task. The injured were treated in many centres throughout the country. In our hospital, all relevant units provided multidisciplinary service to our earthquake victims.

Superficial injuries, fractures, open wounds due to high-energy trauma, compartment syndrome due to compression, and crush injuries are frequently encountered after earthquakes, and patients are usually exposed to multiple traumas. The most common injuries associated with earthquakes are extremity injuries and crush syndrome. First and emergency intervention, including basic life, is usually performed in the disaster area. Emergency surgical procedures such as amputation and fasciatomy may be required for patients with compartment syndrome. The planning of all these surgeries and the follow-up and evaluation of patients require a multidisciplinary approach.

In this study, we planned to retrospectively investigate the anaesthesia management in emergency fasciatomy and amputation surgeries performed in the orthopaedic operating room of patients who were transferred to or admitted to the 3rd level City Hospital during the earthquake disaster on 6 February. We found that anaesthesia data on earthquake victims in the literature were insufficient. We aimed to share our experiences in order to provide guidance in terms of anaesthesia management in possible future disasters.

ELIGIBILITY:
Inclusion Criteria:

* 6 February 2023 earthquake victims who applied to our clinic within 2 months after the earthquake and received anaesthesia and underwent emergency fasciotomy and amputation in the orthopaedic operating room, regardless of gender, aged 18 years and over.

Exclusion Criteria:

* Patients who are not earthquake survivors and under 18 years of age and who have undergone surgery other than fasciatomy or amputation will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age and over who applied to our clinic and received anaesthesia within 2 months after the 6 February 2023 earthquake
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
anaesthetic management in orthopaedic earthquake victims | 2 months (6 February 2023-6 April 2023)
  The effect of general and regional anaesthesia practices of Bilkent City Hospital orthopaedic anaesthesia practitioners on participant prognosis

SECONDARY OUTCOMES:
Metabolic and inflammatory markers | preoperative and postoperative
  Blood levels of CRP, creatine kinase, myoglobin, urea, creatine, haemoglobin, platelets, white blood cells, lymphocytes, inflammation markers,

CONTACTS AND LOCATIONS:
Overall Officials: LEVENT ÖZTÜRK, MD, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No